CLINICAL TRIAL: NCT00763880
Title: Hematoma Blocks in Forearm Fractures: An Effective Adjunct to Procedural Sedation?
Brief Title: Hematoma Block as an Adjunct to Procedural Sedation for Forearm Fracture Reduction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was taking longer than originally anticipated.
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Erika Constantine, Clinical Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CMTT # 4040-05
Record Dates: First submitted 2008-09-26; First posted 2008-10-01 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Forearm Fracture
Keywords: Hematoma block; Lidocaine; Forearm fracture; Radius fracture; Ulna fracture; Ketamine; Midazolam; Procedural sedation
MeSH Terms: conditions — Radius Fractures; Ulna Fractures | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Subjects randomly assigned to this arm will receive 2% lidocaine by injection into their fracture site in the form of a hematoma block.
  Interventions: Drug: Lidocaine
- Normal Saline (Placebo Comparator): Subjects randomly assigned to this arm will receive normal saline by injection into their fracture site
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — 2% Lidocaine (no epinephrine) in the dose of 2.5 mg/kg to a maximum of 10mL will be instilled once into the fracture site in the form of a hematoma block.
  Other Names: Xylocaine; Lidocaine hydrochloride
  Arms: Lidocaine
Drug: Saline — Volume of normal saline equivalent to providing 2.5mg/kg of 2% lidocaine, to a maximum of 10mL.
  Other Names: Sodium Chloride
  Arms: Normal Saline

SUMMARY:
The purpose of our study is to determine if the use of a hematoma block together with intravenous sedation and analgesia is an effective means of managing forearm fractures in the Emergency Department. To determine this, we have designed a randomized, double-blind, placebo controlled trial of hematoma block versus saline for the manipulation of forearm fractures under conscious sedation with ketamine and midazolam. Our hypotheses are two-fold: First, the use of a hematoma block together with conscious sedation will allow for improved pain control. Second, the use of a hematoma block together with conscious sedation will allow us to use less sedation, therefore promoting faster recovery from sedation and more efficient patient turnover in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Ages 3-17
* Closed distal forearm fracture requiring reduction under sedation in the Emergency Department
* Fracture involves the distal third of the forearm

Exclusion Criteria:

* Multiple trauma victims
* Associated nerve or vascular damage
* Associated elbow or humerus injury
* Sensitivity or allergy to lidocaine
* Contraindications to procedural sedation
* Previous attempts at reduction for the same injury

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Total sedation time | Evaluated upon completion of procedure

SECONDARY OUTCOMES:
Non-union | 1 month
Need for re-manipulation | 1 week
Adverse effects of sedation | For the duration of the procedure
Adverse effects of hematoma block | 1 month
Pain control | For entire duration of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Erika Constantine, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital/Rhode Island Hospital, Providence, Rhode Island, United States